CLINICAL TRIAL: NCT06062290
Title: Original Title: Does ElecTromyography Improve preCision and Reliability of nEuromuscular moniToring in paEdiatRic pAtients - A Monocentric Randomized Prospective Agreement Study - ETCETERA
Brief Title: Does Electromyography Improve Precision and Reliability of Neuromuscular Monitoring in Paediatric Patients
Acronym: ETCETERA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Ulm (Other)
Responsible Party: Principal Investigator, Flora Scheffenbichler, Principal Investigator, University Hospital Ulm
Other Study IDs: ETCETERA
Record Dates: First submitted 2023-08-15; First posted 2023-10-02 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Neuromuscular Blockade, Residual; Postoperative Complications
Keywords: Electromyography; Neuromuscular Blockade; Postoperative Complications
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Postoperative Complications | interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- neonates: birth to <28 days
  Interventions: Device: Electromyography (EMG); Device: Kinemyography (KMG)
- infants: 28 days to ≤3 months
  Interventions: Device: Electromyography (EMG); Device: Kinemyography (KMG)
- toddlers: >3 months to ≤2 years
  Interventions: Device: Electromyography (EMG); Device: Kinemyography (KMG)
- children: >2 years to <5 years
  Interventions: Device: Electromyography (EMG); Device: Kinemyography (KMG)

INTERVENTIONS:
Device: Electromyography (EMG) — Measurement of the compound muscle action potential for the assessment of neuromuscular function
Device: Kinemyography (KMG) — Measurement of the muscle velocity for the assessment of neuromuscular function

SUMMARY:
Neuromuscular monitoring is used as a standard surveillance method of neuromuscular function to ensure full recovery at the end of anaesthesia. The currently available devices properly provide respective information in adults but not in children. Furthermore, response to neuromuscular blocking agents differs between adults and children due to age-related differences in body composition, physiological function, and acetylcholine receptor density.

Recently, electromyographic (EMG) technologies to monitor neuromuscular function were increasingly developed including disposables for nerve stimulation and measurement of the compound muscle action potential in children. However, it is still unclear whether the precision and reliability of these devices is superior to the currently available neuromuscular monitoring for children based on kinemyography (KMG).

The ETCETERA study will test the hypothesis that neither EMG nor KMG provides inferior train-of-four readings to the respective reference method in infants and children below five years.

DETAILED DESCRIPTION:
The ETCETERA trial is a randomized clinical agreement study which will prospectively enrol sixty-four children below five years of age scheduled for elective, non-cardiac surgery requiring general anaesthesia and neuromuscular blockade for optimisation of surgical conditions.

The children's neuromuscular function is measured on one hand with EMG and on the other hand with KMG in a randomised fashion. Additionally, randomisation will be stratified upon age groups: 1) neonates: birth to <28 days, 2) infants 28 days to ≤3 months, 3) toddlers: >3 months to ≤2 years, 4) children >2 years to <5 years.

Based on the high failure rate of currently available neuromuscular monitoring devices in infants and neonates, in this randomised agreement study we will primarily compare precision and reliability of EMG and KMG-measured Train-of-Four (TOF) values during spontaneous recovery from a rocuronium-induced neuromuscular blockade in neonates, infants, toddlers, and children <5 years using the age-appropriate paediatric sensors.

ELIGIBILITY:
Inclusion Criteria:

* children and infants < 5 years
* non-cardiac surgery requiring general anaesthesia and neuromuscular blockade
* signed informed written consent
* American Society of Anesthesiologists physical status <4
* intraoperative positioning with access to both arms

Exclusion Criteria:

* allergy to neuromuscular blocking agents
* allergy to neuromuscular monitoring adhesive electrode
* neurologic disease
* surgical procedures outside the operating room
* children receiving neuromuscular blocking agents immediately before surgery

Ages: 1 Hour to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The ETCETERA study will be performed in children <5 years of age scheduled for elective, non-cardiac surgery requiring general anaesthesia and neuromuscular blockade.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Precision of TOF (train of four) measurements | intraoperatively
  The primary endpoint is the repeatability coefficient "r" defined as 1.96 times the standard deviation of the differences between two consecutive TOF ratio measurements on the same patient under identical conditions.
  The repeatability coefficient and its confidence intervals will be calculated using a linear mixed regression model for EMG and KMG measured TOF ratios independently at baseline and at complete neuromuscular recovery, i.e., at TOF ratio > 0.9 and compared between techniques using F-tests with a non-inferiority approach.

SECONDARY OUTCOMES:
Agreement of TOF values during spontaneous recovery of neuromuscular function | intraoperatively
  Agreement of TOF during spontaneous recovery of neuromuscular function, agreement of TOF at baseline and agreement of the final TOF at >0.9 and 1.0 will be verified.
  The repeatability coefficient and its confidence intervals will be calculated using a linear mixed regression model for EMG and KMG measured TOF ratios independently at baseline and at complete neuromuscular recovery, i.e., at TOF ratio > 0.9 and compared between techniques using F-tests with a non-inferiority approach.

OTHER OUTCOMES:
Tactile TOF-count measurement | intraoperatively
  Tactile measurement of TOF response (EMG and KMG)
Postoperative pulmonary events | on the day of surgery in the recovery room
  Including upper airway obstruction, hypoxemia, respiratory distress, aspiration, reintubation (Murphy et al.)
Skin lesions, redness and pressure points on the forearms | on the day of surgery in the recovery room and at hospital discharge or on postoperative day 7, whichever occurs earlier
  Clinical safety outcome
Pain associated with the EMG and KMG measurement | on the day of surgery in the recovery room and at hospital discharge or on postoperative day 7, whichever occurs earlier
  Assessment through child discomfort and pain scale (KUSS) (Bittner et al.)

CONTACTS AND LOCATIONS:
Overall Officials: Flora Scheffenbichler, MD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, University of Ulm, Ulm, Germany.
Locations (1):
- University Hospital Ulm, Ulm, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Buttner W, Finke W, Hilleke M, Reckert S, Vsianska L, Brambrink A. [Development of an observational scale for assessment of postoperative pain in infants]. Anasthesiol Intensivmed Notfallmed Schmerzther. 1998 Jun;33(6):353-61. doi: 10.1055/s-2007-994263. German. PMID 9689392
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT06062290/SAP_000.pdf